CLINICAL TRIAL: NCT00769561
Title: Comparison of a Biofeedback-Based Cognitive Behavioral Treatment and Occlusal Splint Therapy for Temporomandibular Disorders. A Randomized Clinical Trial.
Brief Title: Biofeedback-Based Cognitive Behavioral Treatment for Temporomandibular Disorders
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Philipps University Marburg (Other)
Collaborators: Psychotherapie-Ambulanz Marburg e.V. (Other)
Responsible Party: Principal Investigator, Winfried Rief, PhD, Philipps University Marburg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TMD_Jue2008
Record Dates: First submitted 2008-10-08; First posted 2008-10-09 (Estimated); Results first posted 2013-12-30 (Estimated); Last update posted 2013-12-30 (Estimated); Status verified 2013-12

CONDITIONS: Temporomandibular Disorders
Keywords: Temporomandibular disorders; Biofeedback; Cognitive behavioral therapy; Pain
MeSH Terms: conditions — Temporomandibular Joint Disorders; Pain | interventions — Dental Care; Occlusal Splints

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BFB-CBT (Experimental): Biofeedback-based cognitive-behavioral treatment:
  The biofeedback-based cognitive behavioral intervention comprises 8 individual sessions, each containing both cognitive behavioral and biofeedback elements. Treatment elements are education about the disorder, biofeedback training aimed at improving proprioceptive awareness and reversing parafunctional habits, relaxation techniques, and stress management. Furthermore patients receive portable biofeedback devices for EMG-biofeedback training during day and nighttime in order to reverse diurnal and nocturnal bruxing habits.
  Interventions: Behavioral: Biofeedback-Based Cognitive Behavioral Treatment
- Occlusal Splint (OS) (Active Comparator): Dental treatment with occlusal splints:
  Maxillary or mandibular occlusal splints are made of hard acrylic after taking impressions of the upper and lower dental arches, face bow registration and recording of centric relation. Splints are adjusted to provide even occlusal contact during jaw closing and chewing, and canine and incisor contact during protrusive movements of the jaw. Patients are instructed to use the splint each night and during day time for a period of 7 weeks. One week after initial insertion of the splint patients are requested to return for adjustment.
  Interventions: Device: Dental treatment with occlusal splint (OS)

INTERVENTIONS:
Behavioral: Biofeedback-Based Cognitive Behavioral Treatment — The biofeedback-based cognitive behavioral intervention comprises 8 individual sessions, each containing both cognitive behavioral and biofeedback elements. Treatment elements are education about the disorder, biofeedback training aimed at improving proprioceptive awareness and reversing parafunctional habits, relaxation techniques, and stress management. Furthermore patients receive portable biofeedback devices for EMG-biofeedback training during day and nighttime in order to reverse diurnal and nocturnal bruxing habits.
  Arms: BFB-CBT
Device: Dental treatment with occlusal splint (OS) — Maxillary or mandibular occlusal splints are made of hard acrylic after taking impressions of the upper and lower dental arches, face bow registration and recording of centric relation. Splints are adjusted to provide even occlusal contact during jaw closing and chewing, and canine and incisor contact during protrusive movements of the jaw. Patients are instructed to use the splint each night and during day time for a period of 7 weeks. One week after initial insertion of the splint patients are requested to return for adjustment.
  Arms: Occlusal Splint (OS)

SUMMARY:
The purpose of this study is to develop and evaluate a biofeedback-based cognitive behavioral treatment for patients with chronic temporomandibular disorders using a randomized controlled design.

DETAILED DESCRIPTION:
The purpose of this study is to develop and evaluate a biofeedback-based cognitive behavioral treatment for temporomandibular disorders using a randomized controlled design. 100 patients suffering from chronic temporomandibular disorder are diagnosed using Research Diagnostic Criteria for Temporomandibular Disorders (RDC/TMD). Subsequently, patients are randomly assigned to either a psychological intervention receiving 8 sessions of biofeedback-based cognitive behavioral treatment or to a dental intervention receiving interocclusal splint therapy.

Assessment takes place at baseline, after treatment approximately 8 weeks later, 3 and 6 months follow up. The effects of the interventions are evaluated in terms of reduction in pain intensity, pain related disability, psychological variables such as somatoform symptoms, depression and pain related cognitive adjustment as well as nocturnal electromyographic (EMG) activity.

Additionally, the study aims at identifying variables that predict treatment outcome. Further analyses include initial changes in treatment motivation and illness perceptions and its influence on treatment success, as well as changes in psychophysiological stress reactivity through treatment.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of painful temporomandibular disorder according to Research Diagnostic Criteria for Temporomandibular Disorders (RDC/TMD)
* symptoms persist at least 3 months
* sufficient language skills

Exclusion Criteria:

* somatic diagnosis that requires defined somatic treatment (e.g. occlusal interference)
* presence of a psychotic disorder
* presence of neurological disorders (e.g. dementia)
* alcohol or substance abuse
* presence of other pain condition of predominant severity

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2008-08; Primary Completion 2010-07 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Winfried Rief, Prof. Dr., Study Chair — Department of Clinical Psychology and Psychotherapy, Philipps University Marburg, Germany; Gaby M Bleichhardt, Dr. (PhD), Study Director — Department of Clinical Psychology and Psychotherapy, Philipps University Marburg, Germany; Meike C Shedden Mora, Dipl. Psych., Principal Investigator — Department of Clinical Psychology and Psychotherapy, Philipps University Marburg, Germany
Locations (2):
- Germany (2):
  - Department of Clinical Psychology and Psychotherapy, Philipps University Marburg, Marburg
  - Department of Oral and Maxillofacial Surgery, Philipps University Marburg Medical Center, Marburg

REFERENCES:
- [Result] Shedden Mora MC, Weber D, Neff A, Rief W. Biofeedback-based cognitive-behavioral treatment compared with occlusal splint for temporomandibular disorder: a randomized controlled trial. Clin J Pain. 2013 Dec;29(12):1057-65. doi: 10.1097/AJP.0b013e3182850559. PMID 23446073
- [Result] Shedden Mora M, Weber D, Borkowski S, Rief W. Nocturnal masseter muscle activity is related to symptoms and somatization in temporomandibular disorders. J Psychosom Res. 2012 Oct;73(4):307-12. doi: 10.1016/j.jpsychores.2012.07.008. Epub 2012 Aug 29. PMID 22980538
- [Result] Shedden Mora, M., Bleichhardt, G., Weber, D., Neff, A., & Rief, W. (2010). Biofeedback bei kraniomandibulären Dysfunktionen. Psychotherapeut, 55(3), 217-224.
- See also: Department of Clinical Psychology and Psychotherapy — http://www.uni-marburg.de/fb04/ag-klin/forschung

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Location: Department of Prosthetic Dentistry and the Department of Oral and Maxillofacial Surgery, Marburg Dental School, Philipps University of Marburg, Germany Patient recruitment and follow-up assessment period: August 2008 to April 2011.
Groups:
- BFB-CBT: Biofeedback-based cognitive.behavioral treatment
- Occlusal Splint: Dental treatment with occlusal splint
Period: Overall Study
Arm/Group | BFB-CBT | Occlusal Splint
Started | 29 | 29
Completed | 26 | 24
Not Completed | 3 | 5
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Lost to Follow-up | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BFB-CBT | Occlusal Splint | Total
Number analyzed (Participants) | 29 | 29 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.3 (13.4) | 34.3 (12.5) | 35.3 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 20 | 45
  Male | 4 | 9 | 13
Region of Enrollment [Number; unit: participants]
  Germany | 29 | 29 | 58

OUTCOME MEASURES:

1. Primary Outcome: Pain Intensity (German Pain Questionnaire; Research Diagnostic Criteria for Temporomandibular Disorders (RDC/TMD))
Description: Characteristic pain intensity (German Pain Questionnaire; Research Diagnostic Criteria for Temporomandibular Disorders (RDC/TMD)):
  Characteristic pain intensity was calculated by averaging ratings of current pain, average pain, and worst pain in the past month on a numeric rating scale from 0 (no pain) to 10 (maximum pain), as recommended by RDC/TMD (range 0 - 10). Higher values indicate higher pain levels.
Time Frame: Pre-Post-Design including 3 assessment points: pre-treatment, post-treatment (after 8 weeks), and 6-month follow up
Population: Intent-to-treat approach (ITT) with the last observation carried forward (LOCF)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BFB-CBT | Occlusal Splint
Number analyzed (Participants) | 29 | 29
units on a scale
  Pre-Treatment pain intensity | 5.40 (1.94) | 5.53 (1.97)
  Post-Treatment pain intensity (after 8 weeks) | 3.90 (2.19) | 3.89 (2.40)
  6-months follow up pain intensity | 3.62 (2.48) | 4.21 (2.50)

2. Primary Outcome: Pain Disability (Pain Disability Index)
Description: Pain related disability was assessed using the Pain Disability Index (PDI). The PDI is a brief self-rating scale which assesses the level of pain related disability in seven areas of daily life (e.g., social activity, self-care) on a 0 (no disability) -10 (maximum disability) numeric rating scale (range 0 - 70). Higher values indicate higher disability levels. Cronbach's alpha was .87 in the current sample.
Time Frame: Pre-Post-Design including 3 assessment points: pre-treatment, post-treatment (after 8 weeks), and 6-month follow up
Population: Intent-to-treat approach (ITT) with the last observation carried forward (LOCF)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BFB-CBT | Occlusal Splint
Number analyzed (Participants) | 29 | 29
units on a scale
  Pre-Treatment pain disability | 17.67 (12.75) | 13.88 (13.18)
  Post-Treatment pain disability (after 8 weeks) | 11.07 (12.01) | 11.62 (12.26)
  6-months follow up pain disability | 13.24 (11.96) | 11.61 (11.91)

3. Secondary Outcome: Somatoform Symptoms (Screening for Somatoform Disorders, SOMS)
Description: Somatoform complaints during the past week were assessed using the Screening for Somatoform Symptoms (SOMS-7). 32 medically unexplained symptoms (29 for male subjects) representing DSM-IV criteria for somatization disorder were rated on a 0 ('not at all') to 4 ('very much') scale (range 0 - 128 for women and 0 - 116 for men). A sum score was calculated with higher scores indicating higher intensity and burden of somatoform complaints. In the current sample, Cronbach's alpha level was α = .88.
Time Frame: Pre-Post-Design including 3 assessment points: pre-treatment, post-treatment (after 8 weeks), and 6-month follow up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BFB-CBT | Occlusal Splint
Number analyzed (Participants) | 29 | 29
units on a scale
  Pre-Treatment Somatoform symptoms | 14.97 (13.63) | 11.81 (7.57)
  Post-Treatment Somatoform symptoms (after 8 weeks) | 10.64 (10.16) | 11.30 (9.67)
  6-months follow up Somatoform symptoms | 10.69 (9.67) | 9.81 (7.91)

4. Secondary Outcome: Depressive Symptoms (Centers for Epidemiologic Studies Depression Scale)
Description: Depressive symptoms were measured using the Centre for Epidemiological Studies Depression scale (CES-D). The CES-D asks for the frequency of 20 symptoms of depression during the past week on a scale ranging from 0 ('less than 1 day') to 3 ('5 to 7 days') (range 0-60). Higher scores indicate more depressive symptoms. It is suitable for use in chronic pain patients as it relies less on physical symptoms of depression than do other measures. Cronbach's alpha level in the current sample was α = .89.
Time Frame: Pre-Post-Design including 3 assessment points: pre-treatment, post-treatment (after 8 weeks), and 6-month follow up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BFB-CBT | Occlusal Splint
Number analyzed (Participants) | 29 | 29
units on a scale
  Pre-Treatment Depressive symptoms | 18.51 (11.72) | 17.38 (8.05)
  Post-Treatment Depressive symptoms (after 8 weeks) | 13.05 (8.88) | 16.09 (8.95)
  6-months follow up Depressive symptoms | 15.05 (11.86) | 16.67 (10.07)

5. Secondary Outcome: General Anxiety Symptoms (GAD-7)
Description: General anxiety symptoms were assessed using the 7-item scale from the Patient Health Questionnaire (GAD-7). The GAD-7 asks for anxiety symptoms during the past month on a 1 ('not at all') to 3 ('more than half of the days') rating scale (range 7-21). Higher scores indicate higher levels of anxiety. Cronbach's alpha level in the current sample was α = .64.
Time Frame: Pre-Post-Design including 3 assessment points: pre-treatment, post-treatment (after 8 weeks), and 6-month follow up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BFB-CBT | Occlusal Splint
Number analyzed (Participants) | 29 | 29
units on a scale
  Pre-treatment anxiety | 15.15 (2.62) | 14.15 (2.35)
  Post-Treatment anxiety (after 8 weeks) | 13.07 (3.44) | 13.33 (3.03)
  6-months follow up anxiety | 12.79 (3.27) | 13.04 (2.92)

6. Secondary Outcome: Pain Coping (FESV)
Description: Cognitive and behavioral pain coping strategies were assessed with Coping Strategies Scale from the German Pain Coping Questionnaire (Fragebogen zur Erfassung der Schmerzverarbeitung, FESV). The scale asks for the use of 24 cognitive (e.g. cognitive restructuring) and behavioral (e.g. use of relaxation techniques) strategies for coping with pain on a scale ranging from 1 ('fully disagree') to 6 ('fully agree') (range 24-144). A sum score was used with higher scores indicating more adaptive coping. Cronbach's alpha level was α = .80.
Time Frame: Pre-Post-Design including 3 assessment points: pre-treatment, post-treatment (after 8 weeks), and 6-month follow up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BFB-CBT | Occlusal Splint
Number analyzed (Participants) | 29 | 29
units on a scale
  Pre-Treatment Pain Coping | 62.15 (14.49) | 59.35 (14.56)
  Post-Treatment Pain Coping (after 8 weeks) | 81.80 (19.86) | 64.69 (20.22)
  6-months follow up Pain Coping | 77.11 (21.04) | 60.13 (18.90)

7. Primary Outcome: Jaw Use Limitations (JDL)
Description: Jaw use limitations were measured using the Jaw Disability List (JDL) from the RDC/TMD. The JDL asks the patient to rate interference with eleven oral activities, for example chewing or talking. We used an 11-point numeric rating scale (from 0 'no limitation' to 10 'maximum limitation') instead of ratings of 'yes' and 'no' (range 0 - 110). Higher values indicate higher levels of jaw use limitations. Cronbach's alpha was .86 in the current sample.
Time Frame: Pre-Post-Design including 3 assessment points: pre-treatment, post-treatment (after 8 weeks), and 6-month follow up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BFB-CBT | Occlusal Splint
Number analyzed (Participants) | 29 | 29
units on a scale
  Pre-Treatment Jaw use limitations | 25.87 (21.29) | 27.04 (16.23)
  Post-Treatment Jaw use limitations (after 8 weeks) | 18.52 (17.94) | 18.77 (14.47)
  6-months follow up Jaw use limitations | 18.39 (16.84) | 18.11 (18.02)

8. Secondary Outcome: TMD Related Symptoms
Description: TMD related symptoms, such as jaw pain, toothache or dizziness, were measured using a 41-item TMD symptom list. Following the SOMS-7 scale, intensity of symptoms experienced during the past week was rated from 0 ('not at all') to 4 ('very high intensity') (range 0 - 164). A sum score was built with higher scores indicating higher intensity of TMD related symptoms. The TMD symptom list has not been evaluated previously; however, large bivariate correlations with somatization (Pearson's r = .79), medium to large correlations with pain intensity (r = .48), and medium correlations with depression (r = .37) and anxiety (r = .27) provide evidence of good convergent and divergent validity. Cronbach's alpha level in the current sample was excellent (α = .93).
Time Frame: Pre-Post-Design including 3 assessment points: pre-treatment, post-treatment, and 6-months follow up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BFB-CBT | Occlusal Splint
Number analyzed (Participants) | 29 | 29
units on a scale
  Pre-Treatment TMD related symptoms | 47.69 (24.12) | 37.44 (17.28)
  Post-Treatment TMD related symptoms (at 8 weeks) | 34.34 (22.53) | 28.15 (11.46)
  6-months follow up TMD related symptoms | 35.97 (23.38) | 28.73 (14.89)

ADVERSE EVENTS:
Arm/Group | BFB-CBT | Occlusal Splint
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/29
Other Adverse Events (participants affected / at risk) | 3/29 | 7/29
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BFB-CBT (N=29) | Occlusal Splint (N=29)
Pain in teeth (Nervous system disorders) | 1 (1) | 1 (1) — Patient reported symptom aggravation, namely pain in teeth.
Jaw pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Patient reported symptom aggravation, namely jaw pain
Limited jaw motion (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) — Patient reported symptom aggravation, namely limited jaw motion
Higher muscle tension (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Patient reported symptom aggravation, namely higher muscle tension
Pain in head and/or back (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) — Patient reported symptom aggravation, namely aggravation of pain in head and/or back
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) — Patient reported symptom aggravation, namely ear pain
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1) — Patient reported aggravation of pre-existing tinnitus

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes